CLINICAL TRIAL: NCT04952987
Title: Dry Eye Management With 3% Diquafosol Before and After Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mun Wai Lee (Other)
Collaborators: Santen Oy (Industry)
Responsible Party: Sponsor-Investigator, Mun Wai Lee, Medical Director, LEC Eye Centre
Organization: LEC Eye Centre (Other)
Other Study IDs: LECDQCAT01
Record Dates: First submitted 2021-05-05; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — diquafosol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Diquafosol — Diquafosol (Diquas) is a P2Y2 receptor agonist which improves mucin and tear secretion
  Other Names: Diquas

SUMMARY:
The objective of this study is to evaluate the efficacy of Diquafosol 3% in the management of dry eyes before and after cataract surgery. Patients with pre-existing dry eyes and planned for cataract surgery will be started on Diquafosol eyedrops prior to surgery and treatment will be continued after cataract surgery. Eligible patients will undergo evaluation of dry eye at baseline and subsequently started on treatment with Diquafosol for the duration of 4 weeks before surgery. Further evaluations will be conducted on the day of surgery and at designated time points during and up to 12 weeks after surgery.

DETAILED DESCRIPTION:
Title: Dry Eye Management with 3% Diquafosol Before and After Cataract Surgery

Setting: LEC Eye Centre, Ipoh, Malaysia

Background: Dry eye disease and cataract are two conditions which have been known to increase in incidence with age. Dry eye disease can also be further exacerbated by cataract surgery. Diquafosol (Diquas) is a P2Y2 receptor agonist which improves mucin and tear secretion and is a 'first in class' therapeutic option which has been shown repeatedly to be efficacious in dry eye management.

Objective: To evaluate the efficacy of Diquafosol for dry eye management in patients with pre-existing dry eye disease before and after cataract surgery

Design: Observational case series in a private ophthalmic health facility

Study Plan: Eligible patients will have treatment with Diquas for 4 weeks prior to undergoing cataract surgery. Preoperative clinical evaluation will include documentation of severity of signs and symptoms of dry eye and this will be carried out at baseline, immediately before surgery and subsequently at Week 4 and Week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Eyes with pre-existing dry eye and visually significant cataract planned for phacoemulsification
2. Patients aged18years or older and in good general health
3. Mild to moderate dry eye; non-visually significant ocular surface disease (NVS-OSD) defined as Corneal Fluorescein Staining (CFS) score of <3 on the Oxford scale
4. Tear break-up time (TBUT) <10 seconds

Exclusion Criteria:

1. Eyes with complications after cataract surgery which require a prolonged course of topical medication
2. Eyes with history of contact lens wear in the previous 3 months
3. Eyes with history of regular use of topical eye drops(except artificial tears) in the previous 6 months
4. Treatment history of dry eye beyond artificial tears
5. Eyes with significant ocular surface disease (defined as CFS score of ≥3 on the Oxford scale)
6. Eyes with lacrimal or eyelid disease or ocular surface infections
7. Any ocular surgery within the prior 6 months
8. Using medications that could affect the dry eye condition (eg, antihistamines, antidepressants, decongestants, anticholinergic drugs or hormone treatment)
9. Allergies to Diquafosol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be selected from a population of patients who have mild to moderate dry eye as well as significant cataract listed for phacoemulsification cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Standard Patient Evaluation of Eye Dryness (SPEED) II questionnaire score | 1 month preop, day of surgery, 1month and 3 months postoperatively
  A validated dry eye questionnaire designed to evaluate eye dryness prior to cataract surgery
Change in Tear Break Up Time | 1 month preop, day of surgery, 1month and 3 months postoperatively
  Measure of time taken for ocular tear film to disperse
Change in Conjunctival and corneal fluorescein staining score | 1 month preop, day of surgery, 1month and 3 months postoperatively
  Fluorescein scoring system based on NEI Grading

SECONDARY OUTCOMES:
Change in uncorrected and best corrected visual acuity | 1 month preop, day of surgery, 1month and 3 months postoperatively
  Uncorrected and best corrected distance and near acuity measured with the Snellen chart

CONTACTS AND LOCATIONS:
Overall Officials: Mun Wai Lee, MD, Principal Investigator — LEC Eye Centre
Locations (1):
- LEC Eye Centre, Ipoh, Perak, Malaysia